CLINICAL TRIAL: NCT07325136
Title: A Phase 1/2 Study of BMS-986525 as Monotherapy and in Combination With Nivolumab in Participants With Relapsed/Refractory Small Cell Lung Cancer
Brief Title: A Study to Assess the Safety and Tolerability of BMS-986525 Alone and in Combination With Nivolumab in Participants With Relapsed/Refractory Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA258-0001; 2025-524090-16 (Other: EU CT Number)
Record Dates: First submitted 2026-01-06; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Small Cell Lung Cancer
Keywords: Extensive stage-small cell lung cancer (ES-SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1A: BMS-986525 Monotherapy Dose Escalation (Experimental)
  Interventions: Drug: BMS-986525
- Part 1B: BMS-986525 Combination with Nivolumab Dose Escalation (Experimental)
  Interventions: Drug: BMS-986525; Drug: Nivolumab
- Part 2A: BMS-986525 Monotherapy Dose Expansion (Experimental)
  Interventions: Drug: BMS-986525
- Part 2B: BMS-986525 Combination with Nivolumab Dose Expansion (Experimental)
  Interventions: Drug: BMS-986525; Drug: Nivolumab

INTERVENTIONS:
Drug: BMS-986525 — Specified dose on specified days
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
  Arms: Part 1B: BMS-986525 Combination with Nivolumab Dose Escalation; Part 2B: BMS-986525 Combination with Nivolumab Dose Expansion

SUMMARY:
The purpose of this study is to assess the safety and tolerability of BMS-986525 alone and in combination with Nivolumab in participants with Relapsed/Refractory Small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria

* Participants must have histologically or cytologically documented relapsed/refractory small cell lung cancer (R/R-SCLC).
* Participants must have received at least 1 platinum-based chemotherapy regimen as per locally approved drug labels and institutional guidelines.
* In countries where standard of care first line systemic treatment includes platinum containing chemotherapy in combination with anti-PD-(L)1 therapy, it is required that participants have progressed on, are ineligible for or not have access to an anti-PD- (L)1 therapy.

Exclusion Criteria

* Participants must not have any untreated CNS metastases.
* Participants must not have an active, known or suspected autoimmune disease.
* Participants must not have had a prior organ or tissue allograft.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-02-18 (Estimated); Primary Completion 2029-04-23 (Estimated); Study Completion 2029-04-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to approximately 2 years
Number of participants with serious adverse events (SAEs) | Up to approximately 2 years
Number of participants with AEs meeting dose-limiting toxicity (DLT) criteria | Up to 21 days
Number of participants with AEs leading to discontinuation | Up to approximately 2 years
Number of participants with AEs leading to death | Up to approximately 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumor Version 1.1 (RECIST v1.1) by investigator assessment | Up to approximately 3 years
Maximum observed concentration within a dosing interval (Cmax) | Up to approximately 2 years
Time of maximum observed plasma concentration within a dosing interval (Tmax) | Up to approximately 2 years
Area under the concentration-time curve within a dosing interval (AUC(TAU)) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- United States (5):
  - Local Institution - 0011, Detroit, Michigan
  - Local Institution - 0026, Buffalo, New York
  - Local Institution - 0005, Durham, North Carolina
  - Local Institution - 0004, Cleveland, Ohio
  - Local Institution - 0006, Nashville, Tennessee
- Local Institution - 0001, Rozzano, Milano, Italy
- Japan (2):
  - Local Institution - 0020, Hirakata, Osaka
  - Local Institution - 0018, Chuo-ku, Tokyo
- Romania (2):
  - Local Institution - 0023, Timișoara, Timiș County
  - Local Institution - 0003, Craiova
- Local Institution - 0009, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com